CLINICAL TRIAL: NCT06363786
Title: Mitigating the Impact of Absorbent Products on Skin Occlusion: Changes to Skin Microbiome and Skin Parameters Due to Reduction of Skin Surface pH in Healthy Participants
Brief Title: Reducing Skin Surface pH During Skin Occlusion: Changes to Skin Microbiome and Skin Parameters
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Essity Hygiene and Health AB (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: GOOSEBERRY
Record Dates: First submitted 2024-04-09; First posted 2024-04-12 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2025-02

CONDITIONS: Incontinence-associated Dermatitis

STUDY DESIGN:
Intervention Model Description: Healthy volunteers get patches carrying a low pH or control formula applied to the forearms. The patches are carried over two days and the skin parameters and skin microbiome is measured on day 3.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Test patches (Experimental): Application of test patches. Each subject wear both low pH formula patches (intervention) and control patches without formula.
  Interventions: Other: Test patches

INTERVENTIONS:
Other: Test patches — Patches (incontinence product cut outs) with a low pH formula or control patches without formula.

SUMMARY:
The main aim of this exploratory research study is to investigate how exposure to a material with low pH affects the skin microbiome and skin parameters. This investigation involves an experimental setup in which application of test patches with lowered pH levels or control patches without lowered pH are used. The test patches are applied on healthy adult volunteers. About 20 subjects are planned for the study. The skin microbiome preservation and diversity will be addressed employing Molecular Sequencing and quantitative polymerase chain reaction (qPCR). In addition, skin pH, composition and hydration will be measured with various methods, e.g., AquaFlux, Moisture Meter, TEWL and Confocal Raman spectroscopy. The study will span three consecutive days in total. Each participant will be provided with four patches on each forearm: two patches will be applied to each dorsal forearm and two on each volar forearm. The first day will be for study inclusion and application of patches. In day two the patches will be changed and on day three measurements for pH, TEWL, skin hydration, Raman and tape stripping will be conducted and sampling for Molecular Sequencing and qPCR measurements will be done. There is no formal hypothesis in the study but our idea is that utilizing patches with a lower pH could maintain the diversity and richness of the natural skin microbiome while retaining and even enhancing key skin barrier parameters. A descriptive analysis will be conducted for all measurements with appropriate statistical tests on 5% level for variables. In addition to descriptive data analysis statistics, Clinical Microbiomics and Bio-Me Microbiome Profiling will employ various statistical methods, such as paired Mann-Whitney U tests. The Benjamini-Hochberg (BH) method to control the false discovery rate (FDR) will be employed.

ELIGIBILITY:
Inclusion Criteria:

1. Signed Informed Consent Form
2. Male and female ≥18 and ≤80 years.
3. Willingness and ability to comply with study procedures, visit schedules, and requirements.
4. Intact skin on the forearms without any signs of irritation.
5. Agree not to shower or use cosmetic products on the arms the day before visit 1 and during the study period.
6. Agree not to engage in intense physical activity throughout the study period.

Exclusion Criteria:

1. Have any known allergies or intolerances to one or several components of the absorbing incontinence/menstrual products.
2. Have any known allergies or intolerances to one or several ingredients in cosmetic products.
3. Have an ongoing skin irritation/infection on the forearms.
4. Have any skin conditions such as psoriasis and eczema.
5. Have any tattoos on the forearms.
6. Suffer from excessive sweating, hyperhidrosis.
7. Have immunodeficiency or any other condition that makes participation in the clinical investigation inappropriate, as judged by investigator.
8. Have an alcohol and/or drug dependency.
9. Have had active sunbathing on arms latest 2 weeks prior to study.
10. Have used tanning or bleaching products on arms at least 1 month before the study starts.
11. Have performed hair removal on the arms 1 month prior to the study.
12. Are pregnant or nursing.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2024-04-15 (Actual); Primary Completion 2024-05-30 (Actual); Study Completion 2024-08-30 (Actual)

PRIMARY OUTCOMES:
Changes in skin microbiome as measured by molecular sequencing | 2 days
  Molecular sequencing is used to provide taxonomic insight and overview of microbial diversity on the skin. Skin under the test and control patches are compared.
Changes in skin microbiome diversity as measured by qPCR | 2 days
  qPCR is employed to analyse and quantify specific microbial species or groups. Skin under the test and control patches are compared.
Skin surface pH | 2 days
  The change in skin surface pH under the test and control patches are compared.

SECONDARY OUTCOMES:
Change in Trans Epidermal Water loss | 2 days
  As measured by Dermalab instrument. Transepidermal water loss (TEWL) as measured under the test and control patches.
Change in skin hydration | 2 days
  Skin hydration (SH) as measured with moisture meter instrument under the test and control patches.
Change in Skin water profile | 2 days
  As measured Confocal raman microspectrometry. The water content of skin at different depths is measured and compared for the skin under test and control patches.
Presence of low pH formula on the skin | 2 days
  The extent on formula transfer to the skin as measured with tape stripping.

CONTACTS AND LOCATIONS:
Overall Officials: Ulrika Husmark, PhD, Principal Investigator — Essity Hygiene and Health AB
Locations (1):
- Essity Study Site, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: No